CLINICAL TRIAL: NCT01853514
Title: Assessing Consumer Behavior Regarding the Purchasing of Fresh Produce in Low-income Population
Brief Title: Fresh Fruit and Vegetable Purchasing Behavior
Status: Completed | Type: Observational
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Responsible Party: Sponsor
Other Study IDs: 2013-020
Record Dates: First submitted 2013-05-03; First posted 2013-05-15 (Estimated); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Low-income Population
Keywords: Low income; Fruit and vegetables; Conventional produce; Organic produce; Pesticide; Purchasing behavior; Message framing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Low income: Income level equal or less than 250% above the poverty level

SUMMARY:
Primary objective is to determine the impact of messages related to conventionally grown and organically grown produce on purchasing behaviors in low-income individuals.

Secondary objective is to assess knowledge and attitudes about conventionally and organically grown fruit and vegetable in low-income individuals.

DETAILED DESCRIPTION:
This is a cross-sectional study that will evaluate consumer behavior related to the purchasing of fresh produce in the low-income population through a self-report survey questionnaire.

A sample size of 500 subjects is planned. A screening questionnaire will be provided to each subject to determine their eligibility to be in the study. The screening questionnaire consists of 6 questions related to household income level, grocery shopping frequency, employment field, and age. For subjects who are determined to be eligible, they will be asked to complete the study survey questionnaire.

The survey questionnaire consists of 53 questions to assess subject's beliefs and knowledge about organic and conventional fresh fruits and vegetables and how their beliefs and knowledge affect their purchasing behavior related to organic and conventional fresh produce. There are five major categories in the survey to assess different dimensions that influence subjects' purchasing decisions regarding fresh produce. The categories are issue awareness, purchasing behavior, message framing, credibility, and demographics. Issue awareness is used to assess the subjects' previous knowledge, beliefs and attitude towards organic and conventional fresh produce. Purchasing behavior is used to understand why subjects purchase organic or conventional fresh produce. Message framing is used to determine whether message framing has an impact on the self-reported likelihood to purchase organic or conventional fresh produce. Credibility is used to find which source subjects trust the most regarding fresh produce information. Lastly, demographic information will be obtained to analyze characteristic differences.

ELIGIBILITY:
Inclusion Criteria:

* Low income equal or less than 250% above the poverty level.
* 18 years of age and older
* People who do some or most grocery shopping

Exclusion Criteria:

* Employment in any of the following fields: Print, Online/Broadcast Media, Market Research, Advertising, Health, Nutrition, Public Relations
* Rarely or never purchases groceries
* Does not meet low-income qualification criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Low income equal or less than 250% above the poverty level.
Sampling Method: Probability Sample
Enrollment: 510 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2013-01-09 (Actual); Study Completion 2013-01-09 (Actual)

PRIMARY OUTCOMES:
Data collection on Change in likelihood on reported purchasing behavior, as measured by questionnaire, on conventional and organic fresh fruits and vegetables prior and after message testing | 1 hr
  purchasing behavior, as measured by questionnaire, on conventional and organic fresh fruits and vegetables prior and after message testing

SECONDARY OUTCOMES:
Data collection on Effect of issue awareness, attitude, and knowledge related to conventional and organic fresh fruits and vegetables, as measured by questionnaire, on fresh produce purchasing behaviors prior message testing. | 1 hr
  issue awareness, attitude, and knowledge related to conventional and organic fresh fruits and vegetables, as measured by questionnaire, on fresh produce purchasing behaviors prior message testing

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, Ph.D, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided